CLINICAL TRIAL: NCT01680614
Title: The Efficacy of Computerized Alcohol Screening and Intervention (CASI) in At-Risk Emergency Department and Trauma Patients
Acronym: CASI
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Shahram Lotfipour, Principal Investigator, University of California, Irvine
Other Study IDs: 2011-8155
Record Dates: First submitted 2012-09-04; First posted 2012-09-07 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Alcohol Consumption
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- At Risk Adult Drinkers: CASI
  Interventions: Behavioral: CASI

INTERVENTIONS:
Behavioral: CASI

SUMMARY:
The purpose of this research is to examine the effectiveness of computerized alcohol screening and brief intervention in the UC Irvine Medical Center Emergency Department (ED) and Trauma Patients. Brief interventions have a high potential impact in ED and Trauma populations. Computerized alcohol screening and brief intervention (CASI) is a fast and easy to use tool for patients and healthcare providers. CASI mitigates barriers to proper screening and intervention, including time, availability of trained personnel, patient comfort, and language barriers. CASI provides the Alcohol Use Disorders Identification Test (AUDIT) followed by a brief intervention and customized alcohol intake recomendations for the patient.

The intervention of this study will be the addition of a brief CASI questionnaire to the standard of care for a random subset of subjects. All subjects who screen positive for hazardous alcohol use will be followed up and reassessed for alcohol use. The researchers hypothesize that the addition of CASI will lead to a decrease in alcohol intake within three months. The basis of this research is evidence of the effectiveness in the CASI system, the growing public health issue of alcohol abuse, the need to be able to provide effective screening and brief intervention in the high volume ED settings, and findings that the primary method to reduce traumatic death is prevention.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Trauma and ED patients

Exclusion Criteria:

* Under the age of 18
* Intoxicated
* Psychiatric

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Emergency Department
Sampling Method: Probability Sample
Enrollment: 2114 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2015-06-01 (Actual); Study Completion 2015-06-29

CONTACTS AND LOCATIONS:
Locations (1):
- UC Irvine Medical Center, Orange, California, United States

REFERENCES:
- See also: Center for Trauma and Injury Prevention Research — http://www.ctipr.uci.edu